CLINICAL TRIAL: NCT03308461
Title: Fecal Microbiota Transplantation for Constipation With Difficult Defecation
Brief Title: Fecal Microbiota Transplantation for Constipation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Faming Zhang, Associate professor, Gastroenterology, The Second Hospital of Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMT-CN-160107
Record Dates: First submitted 2017-10-07; First posted 2017-10-12 (Actual); Last update posted 2017-10-12 (Actual); Status verified 2016-05

CONDITIONS: Gut Microbiota; Constipation
Keywords: difficult defecation; fecal microbiota transplantation; stool pattern
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fecal microbiota transplantation (FMT) (Experimental): Patients underwent single FMT in this studyAll patients were assessed before FMT and during 12-week follow-up after FMT.
  Interventions: Drug: Fecal Microbiota suspension

INTERVENTIONS:
Drug: Fecal Microbiota suspension — The prepared microbiota suspension was infused into mid-gut.

SUMMARY:
Difficult defecation is a common symptom involving with patients'life quality. The stool pattern of these patients might be related to the contribution of gut microbiota. This pilot study proposed hypothesis that stool pattern could be used as a simple index to screen the potential candidates of fecal microbiota transplantation in patients with difficult defecation.

DETAILED DESCRIPTION:
Difficult defecation is a common symptom involving with patients'life quality. The stool pattern of these patients might be related to the contribution of gut microbiota. This pilot study proposed hypothesis that stool pattern could be used as a simple index to screen the potential candidates of fecal microbiota transplantation in patients with difficult defecation. Patients underwent single FMT in this study were divided into hard-stool group and loose-stool group. All patients were assessed before FMT and during 12-week follow-up after FMT.

ELIGIBILITY:
Inclusion Criteria:

1. age between 14-80 years old;
2. difficult defecation with more than six months (a. straining during defecation; b. sensation of incomplete evacuation; c. sensation of anorectal blockage; d. manual maneuvers to facilitate defecation).

Exclusion Criteria:

1. difficult defecation due to secondary factors (e.g. drugs, pelvic surgery, psychiatric disorders);
2. with history of gastrointestinal diseases such as cancer, inflammatory bowel diseases (IBD);
3. pregnant or breast-feeding women;
4. infection with pathogenic bacteria. Enrolled patients were divided into hard-stool group and loose-stool group according to their stool patterns. All patients were followed up for 12 weeks.

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-05-01 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
defecation frequency | 12 weeks
  frequency of defecation per week
stool consistency | 12 weeks
  The category of stool consistency score based on the BSS (Bristol Stool Form Scale)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Center for Digestive Diseases, The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Vandeputte D, Falony G, Vieira-Silva S, Tito RY, Joossens M, Raes J. Stool consistency is strongly associated with gut microbiota richness and composition, enterotypes and bacterial growth rates. Gut. 2016 Jan;65(1):57-62. doi: 10.1136/gutjnl-2015-309618. Epub 2015 Jun 11. PMID 26069274
- [Background] Tigchelaar EF, Bonder MJ, Jankipersadsing SA, Fu J, Wijmenga C, Zhernakova A. Gut microbiota composition associated with stool consistency. Gut. 2016 Mar;65(3):540-2. doi: 10.1136/gutjnl-2015-310328. Epub 2015 Aug 14. No abstract available. PMID 26276682
- [Background] Duncan SH, Louis P, Flint HJ. Lactate-utilizing bacteria, isolated from human feces, that produce butyrate as a major fermentation product. Appl Environ Microbiol. 2004 Oct;70(10):5810-7. doi: 10.1128/AEM.70.10.5810-5817.2004. PMID 15466518